CLINICAL TRIAL: NCT02759445
Title: Detection of Early Changes in Left Ventricular Function by Myocardial Deformation Imaging After Acute Excessive Alcohol Ingestion
Brief Title: Myocardial Deformation Imaging After Acute Alcohol Excess
Acronym: C2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: C2-Strain; 14-110 (Other: CTC-A)
Record Dates: First submitted 2015-11-24; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Myocardial Dysfunction
Keywords: alcohol induced cardiomyopathy; myocardial deformation imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: routine treatment — No intervention, only observation and describing

SUMMARY:
Background: Chronic excessive alcohol consumption leads to progressive and chronic cardiac dysfunction. In general, patients consuming alcohol more than five years are at risk for the development of dilated cardiomyopathy. As only few data about immediate changes in left ventricular function after acute excessive alcohol ingestion are available, this study sought to close this gap.

Methods: 200 subjects (not used to alcohol, no cardiac disease) will be examined up to 12 hours after alcohol excess and after 4 weeks of complete alcohol abstinence. Echocardiography will performed at baseline and at follow-up regarding conventional parameter [as left ventricular ejection fraction (LVEF), transmitral early (E) and late (A) Doppler flow velocities, E/A ratio, deceleration time of E (DT) and isovolumic relaxation time (IVRT)] and myocardial deformation data [as layer specific global circumferential (endo GCS, mid GCS, epi GCS) and longitudinal (endo GLS, mid GLS, epi GLS) strain].

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects who are not used to alcohol
* subjets who had an excessive alcohol Ingestion up to 12 hours before echocardiography

Exclusion Criteria:

* any heart disease
* subjects under 18 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who are not used to alcohol and have no heart disease will be asked for an echocardipgraphy (at baseline and at 4 weeks follow-up) in case of excessive alcohol Ingestion up to 12 hours before determination
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Myocardial Dysfunction by echocardiographic parameters | At 4 weeks follow-up
  Conventional echocardiographic parameters as left ventricular ejection fraction (measured in %) and volumes (measured in ml) and myocardial Deformation parameters as global and layer specific radial, longitudinal and circumferential strain (all measured in %) will be determined

SECONDARY OUTCOMES:
Change from baseline in echocardiographic parameters | from baseline to follow up at 4 weeks
  These echocardiographic parameters will be determined at baseline and at 4 weeks follow up and the changes (assessed by percentage differences) will be given

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, Prof., Principal Investigator — Department of Internal Medicine I, University Hospital Aachen
Locations (1):
- Department of Cardiology, RWTH Aachen University Hospital, Aachen, Germany